CLINICAL TRIAL: NCT00523016
Title: A Pilot Study Investigating the Feasibility of Using Acupuncture Treatment to Reduce Below-Level Neuropathic Pain in Spinal Cord Injury.
Brief Title: Acupuncture Treatment to Reduce Burning Pain in Spinal Cord Injury
Acronym: APSCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of British Columbia (Other)
Responsible Party: Principal Investigator, Linda M. Rapson, Adjunct Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRI REB # 07-045
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Neuropathic Pain
Keywords: acupuncture; electroacupuncture; sham acupuncture; spinal cord injury; neuropathic pain; burning pain
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries; Pain | interventions — Electroacupuncture; Acupuncture Therapy; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroacupuncture (Experimental): Subjects will receive Lyndhurst Central Neuropathic Pain Acupuncture Protocol (LCCNPAP) electroacupuncture protocol for 20 minutes per treatment session; a total of 13 treatments will be administered over 3-4 weeks.
  Interventions: Procedure: Lyndhurst Central Neuropathic Pain Acupuncture Protocol (LCCNPAP)
- Sham acupuncture (Sham Comparator): Subjects will receive simulated acupuncture that includes insertion of acupuncture needles on the head. During each treatment session, needles will be stimulated with electricity for 20 minutes. A total of 13 treatments will be administered over 3-4 weeks. This group will be offered the LCCNPAP treatment at the completion of study participation.
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Lyndhurst Central Neuropathic Pain Acupuncture Protocol (LCCNPAP) — LCCNPAP: acupuncture needle insertion at acupuncture points on the head that will be stimulated with electricity from a battery-operated Chinese acupuncture stimulation device for 20 minutes. A total of 13 treatments will be administered over 3-4 weeks.
  Other Names: Electroacupuncture; Acupuncture + Electrical Stimulation
  Arms: Electroacupuncture
Procedure: Sham acupuncture — Sham acupuncture: Simulated acupuncture that includes insertion of acupuncture needles on the head that will be stimulated with electricity from a battery-operated Chinese acupuncture stimulation device for 20 minutes. A total of 13 treatments will be administered over 3-4 weeks. This group will be offered the LCCNPAP treatment at the completion of study participation.
  Other Names: Placebo acupuncture
  Arms: Sham acupuncture

SUMMARY:
Acupuncture has been used with good results for many years at Toronto Rehabilitation Institute Lyndhurst Centre (Toronto, ON, Canada), Parkwood Hospital (London, ON, Canada) and GF Strong Rehabilitation Institute (Vancouver, BC, Canada) to reduce burning pain in individuals with spinal cord injuries (SCI). This multi-centre RCT will test an acupuncture protocol for treatment of burning pain in 40 people with burning pain in SCI, using a sham acupuncture protocol as the control.

Objectives of Study:

1. To determine the feasibility of conducting a real acupuncture vs. sham acupuncture trial in a multi-centre study using the Lyndhurst Central Neuropathic Pain Acupuncture Protocol (LCCNPAP). This will inform a larger study which will directly evaluate the effect of the LCCNPAP on pain and Quality of Life (QOL) in individuals with SCI.
2. To determine which outcome measures are most responsive and the amount of change that could be expected, with respect to pain and QOL, for the larger study.
3. To obtain preliminary data to determine subject numbers for future studies evaluating the effect of the acupuncture protocol.

DETAILED DESCRIPTION:
40 individuals with SCI below-level neuropathic pain who are at least 6 weeks post-injury will be recruited at the three study sites. Subjects will be randomized into either the experimental or control group using a random number table as they enter the study to determine whether they will undergo the real acupuncture treatment or sham treatment.

A total of 13 treatments will be administered over a maximum of 4 consecutive weeks with an ideal treatment frequency as follows: 5 times per week during weeks one and two; and 3 times per week during week three.

Following all sessions, whether LCCNPAP group or sham, any adverse events such as nausea, fainting, bleeding etc., will be recorded on an adverse effects sheet for each subject. Baseline arterial blood pressure and heart rate will be monitored at four points during each treatment session for both groups.

ELIGIBILITY:
Inclusion Criteria:

* inpatients or outpatients
* over 18 years of age
* traumatic Spinal Cord Injury* (SCI) onset as an adult. *Traumatic SCI for the purposes of this study, is defined as: 'SCI due to sudden forceful impact on the spinal cord with or without bony injury'.This would include: falls, MVAs, hyperextension injuries, penetrating wounds (gunshot, knives), sports injuries, and exclude: tumours, vascular accidents (AVM), demyelinating conditions, infection, and iatrogenic causes.
* major symptom of burning pain below SCI level
* screened as positive for Central Neuropathic Pain by clinical assessment by Site Investigators which includes completing the LANSS Questionnaire
* English-speaking
* capable of giving informed consent
* on stable pain therapy (i.e. no changes in pain medications for 1 week)

Exclusion Criteria:

* systemic illness
* major psychiatric disorders
* scalp lacerations or infections
* hearing or language problems
* history of diabetes or disease that would affect peripheral nerve function
* pregnancy
* serious co-morbidities
* needle phobia
* having undergone Lyndhurst Centre Central Neuropathic Pain Acupuncture Protocol previously
* having had acupuncture in the last 30 days
* treatment involving use of electrical therapy modalities (i.e. Codetron or TENS) in the last 30 days
* seizure disorders, convulsions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-09; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Improvement in burning pain | Baseline, daily and weekly during treatment, end of study plus 1 month follow up

SECONDARY OUTCOMES:
Improvement in Quality of Life measurements | Baseline, end of study plus 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Rapson, MD, Principal Investigator — Toronto Rehabilitation Institute Lyndhurst Centre; Eva Widerström-Noga, PhD, Study Director — University of Miami; Judith Hunter, PhD, Study Director — University of Toronto; Judi Laprade, PhD, Study Director — University of Toronto; John Clement, MD, Study Director — Parkwood Hospital; Patrick Potter, MD, Study Director — Western University, Canada; Nimmi Bharatwal, MD, Study Director — University of Toronto; Andrei Krassioukov, MD, Study Director — University of British Columbia
Locations (3):
- Canada (3):
  - G. F. Strong Rehabilitation Centre, Vancouver, British Columbia
  - Parkwood Hospital, London, Ontario
  - Toronto Rehabilitation Institute Lyndhurst Centre, Toronto, Ontario